CLINICAL TRIAL: NCT01670695
Title: Cohort Study of Patients With IgG4-Related Disease
Brief Title: A Prospective Cohort Study of IgG4RD in China
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Other Study IDs: IgG4RD-Cohort
Record Dates: First submitted 2012-08-16; First posted 2012-08-22 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: IgG4-related Disease
Keywords: IgG4-related disease; IgG4-RD
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples (serum and plasma, with DNA)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IgG4-RD: Patients with IgG4-RD, including sclerosing pancreatitis, sclerosing cholangitis, inflammatory pseudotumors, retroperitoneal or mediastinal fibrosis, interstitial nephritis, hypophysitis, sclerosing dacryoadenitis, sialadenitis (Mikulicz disease and Küttner's tumor), inflammatory aortic aneurysm, lymphadenopathy, or other inflammatory conditions.

SUMMARY:
This is an cohort study to investigate the disease course and treatment response of patients with IgG4-related disease.

DETAILED DESCRIPTION:
Immunoglobulin G4-related disease (IgG4-RD) is a recently defined emerging clinical entity characterized by tissue infiltration by IgG4-positive plasma cells, tissue fibrosclerosis and elevated serum IgG4 concentration.

In this study, patients with IgG4-RD will be investigated, including clinical presentation, laboratory findings and imaging study. All patients will be treated by standard care and follow-uped for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-75 years old with informed consent
* Patients with IgG4-RD:

  1. swelling, sclerosing and inflammatory involvement of one or more organ, including sclerosing pancreatitis, sclerosing cholangitis, inflammatory pseudotumors, retroperitoneal or mediastinal fibrosis, interstitial nephritis, hypophysitis, sclerosing dacryoadenitis, sialadenitis, inflammatory aortic aneurysm, lymphadenopathy, or other inflammatory conditions;
  2. elevated serum IgG4 (>1.35 g/L)
  3. histopathologic features of fibrosis and/or lymphocytic and polyclonal plasma cell infiltration (and IgG4+ plasma cells on immunohistology when performed);
  4. exclusion of other diseases.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Concurrent severe and/or uncontrolled and/or unstable diseases
* Patient with malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed IgG4-related disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Response | 6 months
  Clinical Response is measured by IgG4-RD Responder Index, including organ/site score and serum IgG4 level.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Principal Investigator — Deptment of Rheumatology, Peking Union Medical College Hospital; Fengchun Zhang, Study Chair — Deptment of Rheumatology, Peking Union Medical College Hospital
Locations (1):
- Deptment of Rheumatology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Luo X, Peng Y, Zhang P, Li J, Liu Z, Lu H, Zhang X, Zeng X, Zhang F, Fei Y, Zhang W. Comparison of the Effects of Cyclophosphamide and Mycophenolate Mofetil Treatment Against Immunoglobulin G4-Related Disease: A Retrospective Cohort Study. Front Med (Lausanne). 2020 Jul 7;7:253. doi: 10.3389/fmed.2020.00253. eCollection 2020. PMID 32733900